CLINICAL TRIAL: NCT03449498
Title: The Effects of Intensive Therapy on Quantitative and Qualitative Parameters of Trunk and Lower Limbs in Children With Spastic Cerebral Palsy.
Brief Title: The Effects of Intensive Therapy on Trunk and Lower Limbs in Children With Spastic Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/0678
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Intensive qualitative functional therapy
  Interventions: Other: Qualitative functional therapy
- control group (Experimental): Intensive functional therapy
  Interventions: Other: Functional therapy

INTERVENTIONS:
Other: Qualitative functional therapy — Camps fot children with spastic CP are organised. Each camp consists of 10 days of 6 hours therapy per day. Six functional activities focusing on lower limbs and trunk are performed: walking, stair climbing, balance, transfers, trunk control, and Wii (combination of functional activities in sitting and/or standing). A group of clinical experts composes a set of exercises for each of these activities, however individual adaptations according to the needs and abilities of the child can be still be done. Quality of movement (alignment, weightshift, dissociation, coordination and stability) is hereby very important. The theme 'circus' is used to enhance the motivation of the children.
  Arms: study group
Other: Functional therapy — Camps fot children with spastic CP are organised. Each camp consists of 10 days of 6 hours therapy per day. Goals are set with the parents and the children. During the camp children work on obtaining these goals in a exclusively functional way.
  Arms: control group

SUMMARY:
Research on the effects of physiotherapeutic interventions in children with CP has grown expansively, and shows a wide diversity of techniques and concepts that are used in variable intensity. Until now there is no consensus on the optimal intensity of these interventions to have a positive impact on the activity and participation level of these children. A recent systematic review and meta-analysis already showed evidence for the effect of intensive training of hand function in children with CP, including short bursts of highly intensive therapy. In contrast, studies on the effect of intensive therapy of gross motor function were limited, and training was performed at a lower intensity during a longer period, resulting in effects that are more inconclusive. Moreover, none of the reviewed studies included improvement of trunk control as one of their treatment goals, although it is known that most children with CP experience some problems with trunk control, to a variable extent.

This research project has two aims, i.e. 1) investigating the effect of intensive therapy camps on qualitative and quantitative parameters of lower limbs and trunk; and 2) comparing the effect of two therapeutic approaches, namely a functional approach versus a more qualitative-functional approach on these parameters.

DETAILED DESCRIPTION:
Research on the effects of physiotherapeutic interventions in children with CP has grown expansively, and shows a wide diversity of techniques and concepts that are used in variable intensity. Until now there is no consensus on the optimal intensity of these interventions to have a positive impact on the activity and participation level of these children. A recent systematic review and meta-analysis already showed evidence for the effect of intensive training of hand function in children with CP, including short bursts of highly intensive therapy. In contrast, studies on the effect of intensive therapy of gross motor function were limited, and training was performed at a lower intensity during a longer period, resulting in effects that are more inconclusive. Moreover, none of the reviewed studies included improvement of trunk control as one of their treatment goals, although it is known that most children with CP experience some problems with trunk control, to a variable extent.

This research project has two aims, i.e. 1) investigating the effect of intensive therapy camps on qualitative and quantitative parameters of lower limbs and trunk; and 2) comparing the effect of two therapeutic approaches, namely a functional approach versus a more qualitative-functional approach on these parameters.

ELIGIBILITY:
Inclusion Criteria:

1. spastic type of CP
2. bilateral motor involvement (both diplegia and quadriplegia)
3. GMFCS-level II and III
4. 6 to 12 years old
5. cognition: able to understand and execute instructions in a proper way and sufficient concentration (both during the measurements as during the camp).

Exclusion Criteria:

1. mixed form of CP (with ataxia or dystonia)
2. Botulinum Toxin-A injections within six months prior to the camp
3. multilevel orthopedic surgery within one year prior to the camp
4. selective dorsal rhizotomy within two years prior to the camp
5. spinal fusion

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Quality Function Measurement (QFM) and the Gross Motor Measurement Scale (GMFM) | 1h30
  The Gross Motor Function Measure (GMFM)25 is used for the evaluation of gross motor function. The GMFM-88 exists of 88 items categorized into five dimensions: Lying & Rolling (Dim A), Sitting (Dim B), Crawling & Kneeling (Dim C), Standing (Dim D), and Walking, Running & Jumping (Dim E). The Quality Function Measure (QFM)26 evaluates the quality of execution of the items of Dim D and E of the GMFM. Five attributes are scored separately by use of video scoring: alignment, coordination, weight shift, stability and dissociated movements.
  GMFM: scale ranges fo each item: 0-3 (0 is the minimum score, 3 is the maximum score). There is a total score for all dimensions and a subscore for each dimension, expressed in a percentage. QFM: scale ranges for each qualitative attribute: 0-3 (0 is the minimum score, 3 the maximum score). There is a total score for each qualitative attribute.

SECONDARY OUTCOMES:
3D-motion analysis system movements of lower limbs and trunk during gait | 1h
  3D-movement analysis is used to evaluate lower limb and trunk movements during gait. The children walk barefoot over a 10m walkway at self-selected speed, while marker trajectories on trunk and lower limbs are captured by 12 infrared cameras (VICON system). Spatiotemporal and kinematic parameters will be evaluated.
Range of motion (passive and active) | 10 minutes
  Assessed with a goniometer (degrees) in standardised positions.
Timed Up and Go | 5 minutes
  Assesses dynamic balance and mobility of the child.
1 Minute Walking Test | 5 minutes
  Evaluates walking ability and endurance of the child.
Muscle tone | 10 minutes
  Modified Ashworth Scale, Tardieu Scale. Scale ranges: 0-4 (0 is the maximum score, 4 is the minimum score).
Muscle strength | 10 minutes
  Daniels and Worthingham's Manual Muscle Testing. Scale ranges: 0-5 (0 is the minimum score, 5 is the maximum score).
Trunk Control Measurement Scale | 30 minutes
  Trunk control in sitting is evaluated with the Trunk Control Measurement Scale (TCMS). The TCMS evaluates two prime aspects of trunk control during functional activities: (1) being a stable base for upper and lower limb movements, and (2) being an actively moving body segment. It consists of three subscales: 'static sitting balance', 'selective movement control' and 'dynamic reaching'.
  Scale range: 0-3 (0 is the minimum score, 3 is the maximum score).

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided